CLINICAL TRIAL: NCT03917095
Title: Mesalazine and Compound Glutamin Enema for the Treatment of Ulcerative Colitis Through Colonic Transendoscopic Enteral Tubing: A Multicenter, Randomized, Controlled Trail
Brief Title: The Safety and Efficacy of TET Enema in the Treatment of UC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TET-CN-190408
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Ulcerative Colitis Chronic Mild; Ulcerative Colitis Chronic Moderate
Keywords: Inflammatory Bowel Disease; Transendoscopic Enteral Tubing; Mesalazine; Compound Glutamine
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Glutamine; Mesalamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Mesalazine conventional enema (Active Comparator): Participants undergo the conventional enema of Mesalazine Enemas (4g) for one week.
  Interventions: Drug: Mesalazine
- Mesalazine TET enema (Experimental): Participants undergo the TET enema of Mesalazine Enemas (4g) for one week.
  Interventions: Device: The Colonic Transendoscopic enteral Tubing.; Drug: Mesalazine
- Compound Glutamine conventional enema (Active Comparator): Participants undergo the conventional enema of Compound Glutamine (24 tablets of the drug were dissolved in 50ml normal saline) for one week.
  Interventions: Drug: Glutamine
- Compound Glutamine TET enema (Experimental): Participants undergo the TET enema of Compound Glutamine (24 tablets of the drug were dissolved in 50ml normal saline) for one week.
  Interventions: Device: The Colonic Transendoscopic enteral Tubing.; Drug: Glutamine
- Compound Glutamine and Mesalazine TET enema (Experimental): Participants undergo the TET enema of Mesalazine(4g) and Compound Glutamine (24 tablets of the drug were dissolved in 50ml normal saline) for one week.
  Interventions: Device: The Colonic Transendoscopic enteral Tubing.; Drug: Glutamine; Drug: Mesalazine

INTERVENTIONS:
Device: The Colonic Transendoscopic enteral Tubing. — The medications were infused into the colon through the Colonic Transendoscopic enteral Tubing(TET).
  Arms: Compound Glutamine TET enema; Compound Glutamine and Mesalazine TET enema; Mesalazine TET enema
Drug: Glutamine — The medications were infused into the colon
  Other Names: Glutamine Product
  Arms: Compound Glutamine TET enema; Compound Glutamine and Mesalazine TET enema; Compound Glutamine conventional enema
Drug: Mesalazine — The medications were infused into the colon
  Other Names: Mesalazine Enema Product
  Arms: Compound Glutamine and Mesalazine TET enema; Mesalazine TET enema; Mesalazine conventional enema

SUMMARY:
Colonic Transendoscopic enteral Tubing(TET) is a novel, safe, convenient, and reliable procedure for Fecal Microbiota Transplantation(FMT).This clinical trail aims to evaluate the efficacy and safety of Mesalazine and Compound Glutamine enema in the treatment of Ulcerative Colitis through Colonic TET.

DETAILED DESCRIPTION:
Enema is a conventional treatment for Ulcerative Colitis(UC). Mesalazine is suitable for the patients with mild to moderate UC.But for the UC with extending lesions, the conventional anema with Mesalazine or other medicine can not very effective.Colonic Transendoscopic enteral Tubing(TET) is a novel, safe, convenient, and reliable procedure for Fecal Microbiota Transplantation(FMT).Compared with the conventional enema, which is only used for local administration, the Colonic TET enema can achieve total colonic administration.This study aims to evaluate the efficacy and safety of Colonic TET for UC.Patients in this study will be divided into 5 groups according to certain criteria: the Mesalazine conventional enema group, the Mesalazine TET enema group, the Compound Glutamine conventional enema group, the Compound Glutamine TET enema group, the Mesalazine and Compound Glutamine TET enema group.Each group was given enema for 7 days.The primary outcome measure was the clinical remission efficacy rate in each group. The secondary outcome measure was the safety of TET.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged between 18 and 65
2. Patients with chronic relapsed mild to moderate active Ulcerative Colitis(left semicolon or extending colonic lesions)
3. Patients who can fully understand this study and voluntarily sign an informed consent;
4. Accept re-examination, follow-up examination and specimen retention in time
5. Suitable for colonoscopy and colonic TET;
6. A history of using Mesalazine and Compound Glutamine safely

Exclusion Criteria:

1. Anti-tumor necrosis factor or methotrexate was used within the first 8 weeks
2. Cyclosporine was used within 4 weeks
3. Antibiotics or probiotics was used within 4 weeks
4. Patients with risk of toxic megacolon, colon cancer or atypical hyperplasia found in pathology
5. History of colon surgery
6. Patients with moderate or severe renal impairment ,abnormal liver function,severe hypertension and cerebrovascular accident
7. Accompanied by other serious diseases, such as cancer or AIDS, that may hinder their enrollment or affect their survival
8. Patients with anxiety, depression, mental or legal disabilities
9. History of suspected or proven alcohol/drug abuse
10. Patients with explosive, massive bloody stools and severe illness who cannot tolerate the colonoscopy
11. Patients who are allergic to salicylic acid or aspirin
12. Patients with food allergies
13. Patients who are preparing to become pregnant during the study period
14. Patients considered by the researchers as unsuitable for enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate | 10-days
  The frequency of defecation and hematochezia score were both zero
The effective rate | 10-days
  Part of the total Mayo score was 3 points lower than the baseline

SECONDARY OUTCOMES:
Adverse events | 10-days
  Number of participants with treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, MD,PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Crispino P, Pica R, Unim H, Rivera M, Cassieri C, Zippi M, Paoluzi P. Efficacy of mesalazine or beclomethasone dipropionate enema or their combination in patients with distal active ulcerative colitis. Eur Rev Med Pharmacol Sci. 2015 Aug;19(15):2830-7. PMID 26241537
- [Background] Jeong SY, Im YN, Youm JY, Lee HK, Im SY. l-Glutamine Attenuates DSS-Induced Colitis via Induction of MAPK Phosphatase-1. Nutrients. 2018 Mar 1;10(3):288. doi: 10.3390/nu10030288. PMID 29494494
- [Result] Peng Z, Xiang J, He Z, Zhang T, Xu L, Cui B, Li P, Huang G, Ji G, Nie Y, Wu K, Fan D, Zhang F. Colonic transendoscopic enteral tubing: A novel way of transplanting fecal microbiota. Endosc Int Open. 2016 Jun;4(6):E610-3. doi: 10.1055/s-0042-105205. Epub 2016 Apr 28. PMID 27556065